CLINICAL TRIAL: NCT01833949
Title: This Prospective Longitudinal Cohort Study Included Infertile Women With PCOS Unresponsive to Clomiphene Citrate Treatment, Who Underwent Either Unilateral (ULOD) or Bilateral (BLOD)Laparoscopic Diathermy
Brief Title: Unilateral Laparoscopic Diathermy Adjusted to Ovarian Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KBC Split (Other)
Responsible Party: Principal Investigator, Martina Šunj, dr.med, KBC Split
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBC-2013-HR
Record Dates: First submitted 2013-04-10; First posted 2013-04-17 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: PCOS
Keywords: polycystic ovary syndrome,laparoscopic ovarian drilling
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ULOD arm (N=49) (Active Comparator): Unilateral laparoscopic drilling
  In the ULOD group, we treated the right ovary.The thermal dose of 60 J applied per one cubic centimeter of ovarian volume was calculated from the mean total energy applied on a 10 cm3 ovary (627 J) from three earlier ULOD reports. Ovarian volume had been measured by ultrasound at baseline to determine the total thermal dose to apply on the right ovary. The number of punctures (Np) was also calculated for each patient according to the following formula:
  Np = 627 J / 30 W / 4 s Therefore, patients in the ULOD group differed in the number of punctures and energy received by the right ovary, depending on its volume.
  Interventions: Procedure: Unilateral laparoscopic drilling
- BLOD arm (N=47) (Active Comparator): Bilateral laparoscopic drilling
  In the comparator, BLOD group, all patients received 600 J per ovary (totaling 1200 J) through five punctures at 30 W for 4 s each (5 punctures x 4 s x 30 W = 600 J).
  The ovaries in both groups were cooled after the drilling by irrigating the abdominal cavity with 200-300 mL of physiological saline.
  Interventions: Procedure: Bilateral laparoscopic drilling

INTERVENTIONS:
Procedure: Unilateral laparoscopic drilling — Unilateral laparoscopic drilling with diathermy adjusted to ovarian volume
  Arms: ULOD arm (N=49)
Procedure: Bilateral laparoscopic drilling — Bilateral laparoscopic drilling with fixed doses energy
  Arms: BLOD arm (N=47)

SUMMARY:
The objective of our study was to compare the efficiency of the right ULOD using thermal doses adjusted to ovarian volume (60 J/cm3) with the BLOD method at constant dose and to assess treatment efficiency.

DETAILED DESCRIPTION:
The study included 96 infertile, clomiphene citrate-resistant women with polycystic ovary syndrome (PCOS), who underwent either unilateral or bilateral laparoscopic diathermy at the Clinical Hospital Split, Croatia. PCOS was diagnosed following the Rotterdam consensus criteria. In the ULOD group, we treated the right ovary with thermal dose of 60 J applied per one cubic centimeter of ovarian. In the comparator, BLOD group, all patients received 600 J per ovary. The follow-up period encompassed six menstrual cycles for all subjects.Sample size was based on the test of the primary hypothesis that ULOD treatment would result in a higher ovulation rate than BLOD. In our pilot study in 61 patients, ovulation rates were estimated to 44% in the BLOD arm and 69% in the ULOD arm. Assuming 5% significance and 80% power, we calculated that the minimal sample size for a one-sided test had to be 96 patients.

The aims of our prospective study:

1. Compare the efficiency of the right ULOD using thermal doses adjusted to ovarian volume (60 J/cm3) with the BLOD method at constant dose and to assess treatment efficiency and predict ovulatory response based on clinical parameters (right or left ovary and its volume) and received thermal doses.
2. Evidence the effects of ULOD using thermal doses adjusted to ovarian volume on endocrine (changes in androgen and AMH) and reproductive outcomes (ovulation rate) in clomiphene-resistant women with PCOS.
3. To determine whether unilateral laparoscopic ovarian drilling (ULOD) using thermal doses adjusted to ovarian volume diminishes ovarian reserve less than bilateral LOD (BLOD) using a fixed thermal dose

ELIGIBILITY:
PCOS was diagnosed following the Rotterdam consensus criteria

Inclusion Criteria:

* age between 25 and 35 years,
* BMI<30 kg/m2,
* infertility period 1-3 years,
* normal partner's semen findings,
* LH≥10 or LH:FSH ratio ≥2,
* testosterone >2.5 nmol/L,
* FAI>4,
* normal oral glucose tolerance test (OGTT).

Exclusion Criteria:

* adrenal hyperplasia,
* thyroid disease,
* Cushing's syndrome,
* hyperprolactinemia,
* tumor-related androgen excess

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Ovulation rate | Six menstrual cycles after LOD for each women
  The main output parameter study is the difference in the rate of ovulation after LOD between the groups with respect to the input parameters (anti-Müller hormone AMH [ng / ml], free androgen index (FAI), T [nmol / L],luteinizing hormone (LH) [IU / L], androstenedione A [nmol / L], the number of follicles in both ovaries (AFC), total ovarian volume [cm3], the volume of the right ovary [cm3], the volume of the left ovary [cm3] and received thermal doses)

SECONDARY OUTCOMES:
Pregnancy | Six menstrual cycles after LOD for each women
  The secondary output parameter is the difference in the probability of pregnancy between the two groups, with the input parameters (AFC, total ovarian volume [cm3], the volume of the right ovary [cm3], the volume of the left ovary [cm3] and received thermal doses), during follow-up of patients (first and sixth cycle after LOD).

OTHER OUTCOMES:
Ovarian reserve | Six menstrual cycles after LOD for each women
  The secondary outcome measures were: correlations and differences in values (and changes) measured markers (unilateral / bilateral or ovulation / anovulation). Markers that are considered: AMH [ng / ml], follicle stimulating hormone (FSH) [IU / L], the number of follicles in both ovaries, total ovarian volume [cm3], the volume of the right ovary [cm3], the volume of the left ovary [cm3], FAI, T [nmol / L], LH [IU / L], A [nmol / L], sex hormone-binding globulin (SHBG) [nmol / L], dehydroepiandrosterone sulfate (DEHASO4), [mmol / L],prolactin (PRL), BMI [kg/m2] and years.

CONTACTS AND LOCATIONS:
Overall Officials: Martina MS Šunj, dr.med, Principal Investigator
Locations (1):
- Clinical Hospital Center Split, Split, Dalmatia, Croatia

REFERENCES:
- [Derived] Sunj M, Canic T, Jeroncic A, Karelovic D, Tandara M, Juric S, Palada I. Anti-Mullerian hormone, testosterone and free androgen index following the dose-adjusted unilateral diathermy in women with polycystic ovary syndrome. Eur J Obstet Gynecol Reprod Biol. 2014 Aug;179:163-9. doi: 10.1016/j.ejogrb.2014.05.011. Epub 2014 Jun 2. PMID 24965999
- [Derived] Sunj M, Canic T, Baldani DP, Tandara M, Jeroncic A, Palada I. Does unilateral laparoscopic diathermy adjusted to ovarian volume increase the chances of ovulation in women with polycystic ovary syndrome? Hum Reprod. 2013 Sep;28(9):2417-24. doi: 10.1093/humrep/det273. Epub 2013 Jul 2. PMID 23820423